CLINICAL TRIAL: NCT04194723
Title: Phase II Clinical Study on the Safety and Efficacy of Antireflux Mucosectomy (ARMS) for Treatment of Gastroesophageal Reflux
Brief Title: Antireflux Mucosectomy (ARMS) for Treatment of Gastroesophageal Reflux
Acronym: ARMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan CHIU, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2016.194T
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Gastro Esophageal Reflux
Keywords: Antireflux Mucosectomy; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antireflux Mucosectomy (Experimental): Antireflux mucosectomy targeted at resection of gastric cardia muocsa to induce fibrosis and improve on the flap value over the gastroesophageal junction
  Interventions: Procedure: Antireflux Mucosectomy

INTERVENTIONS:
Procedure: Antireflux Mucosectomy — ARMS aimed at resection of mucosa at gastric cardia to induce fibrosis and tighten the gastroesophageal junction and reduce acid reflux

SUMMARY:
This is a phase II clinical study to investigate the safety and efficacy of endoscopic antireflux mucosectomy (ARMS) for treatment of GERD.

DETAILED DESCRIPTION:
The objective of the study is to establish the clinical efficacy and safety of ARMS for treatment of GERD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with typical symptoms of GERD with symptomatic response to PPI therapy for ≥ 3 months
2. Hill's grade II and III of the gastroesophageal junction
3. One of the following abnormalities in the objective assessment 3.1. Excessive acid exposure at the distal esophagus evidenced by 24 hour pH tests using % total time pH < 4 and / or DeMeester score 3.2. Endoscopic evidence of LA classes A,B,C or D esophagitis 3.3. Defective LES assessed by HRM with resting pressure of < 6mmHg or total length of less than 4cm or abdominal length of less than 2cm

Exclusion Criteria:

1. Age > 70 yrs of < 18 yrs
2. Pregnancy
3. Any type of Hiatus hernia
4. Patients with underlying malignancy
5. ASA above grade III

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Gastro Esophageal Reflux symptoms | 3 months
  GERD symptoms evidence by the improvement in the Gastroesophageal Reflux Quality of Life (QoL) of ≥50% compared to the baseline off Proton Pump Inhibitors (PPI) value 3 months after the procedure

SECONDARY OUTCOMES:
Technical Success | 1 day
  Success in resection of mucosa at cardia by ARMS
24 hour pH study post ARMS | 3 and 12 months
  24 hour pH study
High resolution Manometry | 3 and 12 months
  HRM
Gastroesophageal junction classified by Hill's classification | 3 and 12 months
  endoscopic assessment of Gastroesophageal junction

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Endoscopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided